CLINICAL TRIAL: NCT05529355
Title: An Exploratory Non-randomized Controlled Trial for Effect and Safety of Envafolimab Combined With Recombinant Human Endostartin Injection/S-1 in Second-line Treatment of Advanced Non-small Cell Lung Cancer
Brief Title: Effect and Safety of Envafolimab Combined With Endostar/S-1 in Second-line of Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anhui Chest Hospital (Other)
Responsible Party: Principal Investigator, Guan Maojing, Dr., Anhui Chest Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z-2014-06-2201
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — envafolimab; endostar protein; S 1 (combination); gimeracil; Endostatins; Tegafur

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Envafolimab plus Endostar and S-1 (Experimental): Envafolimab (300 mg subcutaneously each time, using 4-6 cycles), Recombinant Human Endostartin Injection (210 mg, d1-7 pumps, repeat every 3 weeks, using 4-6 cycles), Tegafur,Gimeracil and Oteracil Porassium Capsules (40 mg Bid, take 2 weeks stop for 1 week, use 4-6 cycles)
  Interventions: Drug: Envafolimab plus Endostar and S-1
- Envafolimab plus Endostar (Active Comparator): Envafolimab (300 mg subcutaneously each time, using 4-6 cycles), Recombinant Human Endostartin Injection (210 mg, d1-7 pumps, repeat every 3 weeks, using 4-6 cycles),
  Interventions: Drug: Envafolimab plus Endostar
- Envafolimab plus S-1 (Active Comparator): Envafolimab (300 mg subcutaneously each time, using 4-6 cycles), Tegafur,Gimeracil and Oteracil Porassium Capsules (40 mg Bid, take 2 weeks stop for 1 week, use 4-6 cycles)
  Interventions: Drug: Envafolimab plus S-1

INTERVENTIONS:
Drug: Envafolimab plus Endostar and S-1 — Immunotherapy combined with chemotherapy and anti VEGFR therapy
  Other Names: Envafolimab combined with Recombinant Human Endostatin Injection/Tegafur,Gimeracil and Oteracil Porassium Capsules
  Arms: Envafolimab plus Endostar and S-1
Drug: Envafolimab plus Endostar — Immunotherapy combined with anti VEGFR therapy
  Other Names: Envafolimab combined with Recombinant Human Endostatin Injection
  Arms: Envafolimab plus Endostar
Drug: Envafolimab plus S-1 — Immunotherapy combined with chemotherapy
  Other Names: Envafolimab combined with Tegafur,Gimeracil and Oteracil Porassium Capsules
  Arms: Envafolimab plus S-1

SUMMARY:
The trial was a randomized, open-label, multicenter Phase II study of patients with advanced or metastatic NSCLC who don't harbor driver genes. The aim is to explore the efficacy and safety of Envafolimab Combined With Endostar/S-1 in second-line treatment of advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
Patients with advanced (stage IV. NSCLC), after signing informed consent, are screened to meet the admission requirements. All the candidates are not randomly placed in 3 treatment groups (which treatment regimen the patient chooses is determined by the clinical supervisor on a patient-by-case basis).

ELIGIBILITY:
Inclusion Criteria:

1. All patients are histologically or cytologically confirmed stage IV non-small cell lung cancer. Genetic testing identifies no driver gene mutations.
2. Male or female, age > 18 years, < 75 years.
3. Patients had not received PD-L1 inhibitors in first-line treatment.
4. KPS score ≥ 70 points (ECOG score 0-1 points), the expected survival ≥3 months;
5. No dysfunction of major organs. EcG, liver function, renal function, and blood count tests before treatment are normal or basically normal, but must meet the following experimental results:

   1. Blood routine test:

      Leukocyte WBC≥3.5×109/L; Neutrophil count (ANC) ≥ 1.5×109/L; Platelet (PLT) ≥ 80×109/L;
   2. Blood biochemical test:

Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal values; Alanine aminotransferase (ALT/SGPT) and alanine transaminases (AST/SGOT) ≤ 2.5 times the normal high value (ULN), or ≤ 5 times the upper limit of normal value in patients with liver metastases; Serum creatinine (Cr) ≤ 1.5 times the upper limit of normal values; c. Cardiac function test: 50% of the left ventricular ejection function of the heart >; 6) The subject has good compliance, and can cooperates with follow-up.

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-09-18 (Estimated); Primary Completion 2023-09-18 (Estimated); Study Completion 2023-09-18 (Estimated)

PRIMARY OUTCOMES:
objective response rate(ORR) | six weeks
  proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors
Adverse events | three weeks
  safety

SECONDARY OUTCOMES:
progression-free survival(PFS) | six weeks
  the time from initial treatment to disease progression
overall survival(OS) | six weeks
  the time from initial treatment to death from any cause